CLINICAL TRIAL: NCT04962373
Title: Brief Admission by Self-referral for Adolescents Who Self-harm, at Risk for Suicide. A Qualitative Study to Optimise and Standardise the Intervention
Brief Title: Brief Admission for Adolescents Who Self-harm
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Sofie Westling, Principal Investigator, Region Skane
Other Study IDs: 2020-01840
Record Dates: First submitted 2021-07-04; First posted 2021-07-15 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Self-Harm, Deliberate; Suicide, Attempted; Suicidal; Non-Suicidal Self Injury
MeSH Terms: conditions — Self-Injurious Behavior; Suicide, Attempted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Adolescents: Adolescents with a contract for Brief admission by self-referral
  Interventions: Other: Semi-structured interviews
- Parents: Parents to adolescents with a contract for Brief admission by self-referral
  Interventions: Other: Semi-structured interviews
- Staff: Health care providers who work with adolescents with a contract for Brief admission by self-referral
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Semi-structured interviews — Each participant will attend a 30-60 minute semi-structured interview conducted by the CI

SUMMARY:
There is still no consensus on how to manage suicidal behavior in youth with recurrent self-harm at times when the risk for suicide is imminent (1). Brief Admission (BA) has evolved as a promising crisis intervention for adults with self-harm (2). The characteristics of BA is different from other types of admission, being focused on prevention through increased autonomy and self-care, based on structured and voluntary brief self-referrals to hospital (3). As a result of a randomized controlled trial, BA is since January 2019, continuously offered to adults with self-harm at risk for suicide in Skåne (4). Parallel to this clinical trial, the method has been adapted to work in a psychiatric setting for adolescents. At present 24 adolescents have access to the method in Skåne. Clinical experiences from staff are promising, however, the lived experiences have not been collected in a standardized way.

The aim of the present study is to gather information on how BA in its present, standardized form works for adolescents, their loved ones and staff working at the ward providing BA. This will be done through semi-structured interviews with:

1. Adolescents using BA and their loved ones
2. Staff working at the ward providing BA. Data will be analyzed with qualitative analysis (5, 6). The ultimate aim is to use these results to optimize the current standardized version of BA for adolescents in order to test in a randomized clinical trial.

ELIGIBILITY:
Sample 1:

Inclusion Criteria:

* Adolescents with an active BA contract
* At least 13 years of age.
* Able to consent to study participation through written and oral information.
* Consent from caregivers
* Given consent to participate

Exclusion Criteria:

* Below the age of 13.

Sample 2:

Inclusion Criteria:

* Parents to adolescents with an active BA contract
* At least 18 years of age.
* Able to consent to study participation through written and oral information.
* Given consent to participate

Exclusion Criteria:

* None

Sample 3:

Inclusion Criteria:

* Staff working with adolescents with an active BA contract
* At least 18 years of age.
* Able to consent to study participation through written and oral information.
* Given consent to participate

Exclusion Criteria:

* None

Ages: 13 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescents with an active BA contract, their loved ones who have given informed consent to participate and psychiatric staff working with the adolescents.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Perceived effective components of Brief Admission for adolescents | 60mins
  Qualitative data from interviews
Potential adaptations of the method to better fit adolescents | 60mins
  Qualitative data from interviews
Areas where Brief Admission have the most prominent perceived effects in adolescents | 60mins
  Qualitative data from interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Psykiatri och habilitering, Region Skåne, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
Data is qualitative, transcriptions from interviews. Even if personal identifiers are removed, it is difficult to ensure enough secrecy/privacy for the participants.

REFERENCES:
- [Background] Strand M, von Hausswolff-Juhlin Y. Patient-controlled hospital admission in psychiatry: A systematic review. Nord J Psychiatry. 2015;69(8):574-86. doi: 10.3109/08039488.2015.1025835. Epub 2015 Apr 2. PMID 25832757
- [Background] Westling S, Daukantaite D, Liljedahl SI, Oh Y, Westrin A, Flyckt L, Helleman M. Effect of Brief Admission to Hospital by Self-referral for Individuals Who Self-harm and Are at Risk of Suicide: A Randomized Clinical Trial. JAMA Netw Open. 2019 Jun 5;2(6):e195463. doi: 10.1001/jamanetworkopen.2019.5463. PMID 31173128
- [Background] Lindseth A, Norberg A. A phenomenological hermeneutical method for researching lived experience. Scand J Caring Sci. 2004 Jun;18(2):145-53. doi: 10.1111/j.1471-6712.2004.00258.x. PMID 15147477
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Background] Helleman M, Lundh LG, Liljedahl SI, Daukantaite D, Westling S. Individuals' experiences with brief admission during the implementation of the brief admission skane RCT, a qualitative study. Nord J Psychiatry. 2018 Jul;72(5):380-386. doi: 10.1080/08039488.2018.1467966. Epub 2018 Apr 27. PMID 29703119
- [Background] Lindkvist RM, Landgren K, Liljedahl SI, Daukantaite D, Helleman M, Westling S. Predictable, Collaborative and Safe: Healthcare Provider Experiences of Introducing Brief Admissions by Self-referral for Self-harming and Suicidal Persons with a History of Extensive Psychiatric Inpatient Care. Issues Ment Health Nurs. 2019 Jul;40(7):548-556. doi: 10.1080/01612840.2019.1585497. Epub 2019 May 17. PMID 31099707
- [Background] Lindkvist RM, Westling S, Liljedahl SI, Landgren K. A Brief Breathing Space: Experiences of Brief Admission by Self-Referral for Self-Harming and Suicidal Individuals with a History of Extensive Psychiatric Inpatient Care. Issues Ment Health Nurs. 2021 Feb;42(2):172-182. doi: 10.1080/01612840.2020.1789787. Epub 2020 Aug 7. PMID 32762578